CLINICAL TRIAL: NCT04690309
Title: Human Versus Analogue Insulin in Patients After Pancreatectomy - Open, Prospective, Randomized, Intervention Study.
Brief Title: Human Versus Analogue Insulin in Patients After Pancreatectomy.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polish Society of Diabetology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Polish Society Of Diabetology
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Pancreatogenous Diabetes
Keywords: human insulin; insulin analogues
MeSH Terms: conditions — Insulin Resistance | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with human insulin preparations (Active Comparator): Treatment with human regular insulin administered subcutaneously before breakfast, lunch and supper and with Neutral Protamine Hagedorn insulin (isofane insulin) administered subcutaneously before sleep.
  Interventions: Drug: Treatment with human insulin preparations or treatment with insulin analogues
- Patients treated with insulin analogues (Active Comparator): Treatment with insulin analogues lispro administered subcutaneously before breakfast, lunch and supper and with glargine administered subcutaneously before sleep.
  Interventions: Drug: Treatment with human insulin preparations or treatment with insulin analogues

INTERVENTIONS:
Drug: Treatment with human insulin preparations or treatment with insulin analogues — The doses of human insulin preparations and insulin analogues will be matched individually to achieve target values of blood glucose - fasting < 100 mg/dl (5.5 mmol/L) and postprandial < 140 mg/dl (7.8mmol/L)

SUMMARY:
Pancreatectomy is a common treatment modality for both benign and malignant pathologies. One of the most common complications after pancreatectomy is pancreatogenous diabetes mellitus. Yet, insulin remains treatment of choice in patients after pancreatectomy, however there is little evidence on the choice of insulin preparation in patients with diabetes after pancreatectomy. In particular, it is unclear whether human or analogue insulin should be preferred in this group of patients.The aim of the study was to compare human vs analog insulin therapy in patients with diabetes prior to or diabetes developing after pancreatectomy performed due to pancreatic tumor. The study was designed as an open, prospective, randomized, intervention study.All patients provided written comprehensive informed consent. After surgery all patients who underwent total pancreatectomy were treated with insulin, while the patients who had partial pancreatectomy performed were treated with basal insulin when fasting plasma glucose exceeded 140 mg/dl and with prandial insulin when 2-hour postprandial plasma glucose exceeded 180 mg/dl.The patients who required insulin treatment after surgery were randomized with the use of random numbers generator (www.randomizer.org) into two groups: Group 1 - treated with insulin analogues (lispro, glargine), Group 2 - treated with human insulin preparations (regular and NPH insulin).The clinical and metabolic assessment was carried out 3 and 6 months after surgery. The study was approved by Local Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

•Patients with pancreatic tumor confirmed in imaging studies and qualified for surgical treatment

Exclusion Criteria:

•Active psychiatric disease not amenable to treatment and hindering cooperation

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic control in patients treated with human insulin preparations insulin vs insulin analogues. | Change in concentration of glycated hemoglobin from baseline to concentration of glycated hemoglobin 6 months after surgery in patients treated with human insulin and insulin analogues
  Metabolic control in patients treated with human insulin and insulin analogues will be assessed using glycated hemoglobin concentration (mmol/mol)

SECONDARY OUTCOMES:
Metabolic control in patients treated with human insulin preparations insulin vs insulin analogues. | Change in concentration of glycated hemoglobin from baseline to concentration of glycated hemoglobin 3 months after surgery in patients treated with human insulin and insulin analogues
  Metabolic control in patients treated with human insulin and insulin analogues will be assessed using glycated hemoglobin concentration (mmol/mol)

CONTACTS AND LOCATIONS:
Locations (1):
- Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes